CLINICAL TRIAL: NCT02392949
Title: Does Passive Spinal Mobilization Improve Shoulders Strength in Healthy Adults?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, LO CHI NGAI, Mr. Lo Chi Ngai, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HSEARS20140926001
Record Dates: First submitted 2015-02-27; First posted 2015-03-19 (Estimated); Last update posted 2016-06-14 (Estimated); Status verified 2016-06

CONDITIONS: Healthy
Keywords: Spine; mobilization

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental group (Experimental): Passive mobilization on cervical spine
  Interventions: Behavioral: Passive mobilization
- Control (Placebo Comparator): Placebo exercise on arms
  Interventions: Other: Placebo

INTERVENTIONS:
Behavioral: Passive mobilization — An anterior-posterior manual pressure act on the cervical spine of the subject
  Arms: Experimental group
Other: Placebo — The elbows will be put into a 90 deg elevated position and held for 5 secs, then back to resting position
  Arms: Control

SUMMARY:
Previous studies have shown that peripheral muscles weakness or inhibition is related to spinal disorders. Passive mobilization and manipulation are likely to reverse such muscle weakness for patients with spinal pain. The purpose of the study was to assess the effect of spinal mobilization on the maximal muscle strength of the shoulders.

DETAILED DESCRIPTION:
Participants without existing neck pain or shoulder problem will be recruited. Subjects will be screened by 2 investigators independently for shoulder muscle weakness. Weakness is determined by the strength of the other side when one side is remarkably weaker or by comparing with the general strength of the deltoid muscle if both sides are suspected involved.

Suitable participants will undergo shoulder strength testing with a handheld dynamometer. Participants will be divided into the intervention group and the control group randomly. The shoulder strength will be tested by the second, individual blinded assessor.

Subjects in the intervention group will receive passive spinal mobilization at cervical 4-5 segment on the involved side(s); the control group will receive placebo intervention.

Each participant will be tested for 2 times, before and immediately after a C4-5 joint mobilization on the involved side (s).

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults

Exclusion Criteria:

* People with active neck or should pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-04; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Deltoid muscle strength (dynamometer) | 10 minutes after the intervention
  Immediate measure after the intervention by dynamometer
Electromyography (EMG) (signal from deltoid muscle) | 10 minutes after the intervention
  The EMG measure on the signal from deltoid muscle immediately after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Chi Ngai Lo, Master, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No